CLINICAL TRIAL: NCT02774941
Title: Comparison of Vibrating Mesh Nebulizer Versus Jet Nebulizer in the Pediatric Asthma Patient a Randomized Controlled Trial
Brief Title: Comparison of Vibrating Mesh Nebulizer Versus Jet Nebulizer in the Pediatric Asthma Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU 112015-091
Record Dates: First submitted 2016-05-13; First posted 2016-05-17 (Estimated); Results first posted 2020-01-31 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Standard single patient-use small volume JN (AirLife™ Sidestream® High-Efficiency Nebulizer, CareFusion, Yorba Linda, CA)
  Interventions: Device: Jet Nebulizer
- Study (Experimental): Vibrating Mesh Nebulizer (Aerogen® Solo with Ultra adapter, Aerogen Ltd, Galway, Ireland)
  Interventions: Device: Vibrating Mesh Nebulizer

INTERVENTIONS:
Device: Jet Nebulizer — Standard single patient-use small volume JN (AirLife™ Sidestream® High-Efficiency Nebulizer, CareFusion, Yorba Linda, CA)
  Arms: Control
Device: Vibrating Mesh Nebulizer — Vibrating Mesh Nebulizer (Aerogen® Solo with Ultra adapter, Aerogen Ltd, Galway, Ireland)
  Arms: Study

SUMMARY:
The purpose of this study is to compare clinical outcomes related to the current practice of using a jet nebulizer (JN) with aerosol mask (AM) or mouthpiece (MP) versus a vibrating mesh nebulizer (VMN) with a valved-mask (VM) or MP in the treatment of acute moderate to severe asthma in Children's Medical Center Dallas Emergency Department (CMCED).

DETAILED DESCRIPTION:
The purpose of this study is to compare clinical outcomes related to the current practice of using a jet nebulizer (JN) with aerosol mask (AM) or mouthpiece (MP) versus a vibrating mesh nebulizer (VMN) with a valved-mask (VM) or MP in the treatment of acute moderate to severe asthma in Children's Medical Center Dallas Emergency Department (CMCED). The investigators hypothesize that using the combination of a VMN and VM or MP will result in fewer hospital admissions and decrease length of stay in CMCED when compared to the current practice of using a JN and AM or MP.

ELIGIBILITY:
Inclusion Criteria:

2 to 18 year old (up to 19th birthday) otherwise healthy children with primary diagnosis of acute moderate to severe exacerbation of asthma presenting to Children's Medical Center Emergency Department, Dallas

-

Exclusion Criteria:

* Children < 2 years old
* Children with comorbid/complex medical conditions such as: congenital or acquired cardiovascular disease, cystic fibrosis, chronic lung disease (other than asthma), bronchopulmonary dysplasia, airway anomalies (e.g., tracheomalacia) or immunodeficiency syndromes.
* Patients with coexisting medical condition such as pneumonia
* Patients in impending respiratory failure as determined by treating physician
* Patients that have had oral corticosteroids within 24hrs of CMCED admission
* Patients that have had bronchodilator treatment within one hour of CMCED admission

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 220 (Actual)
Dates: Start 2016-08; Primary Completion 2019-03-08 (Actual); Study Completion 2019-03-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Medical Center, Dallas, Texas, United States

REFERENCES:
- [Derived] Moody GB, Luckett PM, Shockley CM, Huang R, Ari A. Clinical Efficacy of Vibrating Mesh and Jet Nebulizers With Different Interfaces in Pediatric Subjects With Asthma. Respir Care. 2020 Oct;65(10):1451-1463. doi: 10.4187/respcare.07538. Epub 2020 Mar 24. PMID 32209712

RESULTS

PARTICIPANT FLOW:
Groups:
- Control - Jet Nebulizer: The control group used our standard single patient-use small volume JN (AirLife™ Sidestream® High-Efficiency Nebulizer, CareFusion, Yorba Linda, CA) operated at 7 L/min per manufacture's guidelines.
- Study - Vibrating Mesh Nebulizer: The study group used a VMN (Aerogen® Solo with Ultra adapter, Aerogen Ltd, Galway, Ireland) that is an electronically powered nebulizer.
Period: Overall Study
Arm/Group | Control - Jet Nebulizer | Study - Vibrating Mesh Nebulizer
Started | 110 | 110
Subjects Excluded | 1 | 2
Completed | 109 | 108
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Population: Two children were excluded who were discharged after an initial decision to admit was made and treated after study procedure ended, and one child was excluded after the diagnosis of pneumonia was made.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control - Jet Nebulizer | Study - Vibrating Mesh Nebulizer | Total
Number analyzed (Participants) | 109 | 108 | 217
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 109 | 108 | 217
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 6.0 [5.0 to 10.0] | 7.0 [5.0 to 9.5] | 7.0 [5.0 to 10.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 73 | 146
  Male | 36 | 35 | 71
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 46 | 42 | 88
  Not Hispanic or Latino | 63 | 66 | 129
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 59 | 62 | 121
  White | 48 | 45 | 93
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 109 | 108 | 217
Moderate Asthma [Count of Participants; unit: Participants] | 63 | 46 | 109
Severe Asthma [Count of Participants; unit: Participants] | 46 | 62 | 108

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Hospitalized
Description: The primary outcome measure is rate of hospitalization between the two treatment groups overall
Time Frame: Within emergency department visit time frame (no more than 12 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | Control - Jet Nebulizer | Study - Vibrating Mesh Nebulizer
Number analyzed (Participants) | 109 | 108
Participants | 22 | 15

2. Secondary Outcome: Number of Treatments Required to Achieve Mild Asthma Score - Discharge Criteria
Time Frame: Within emergency department visit time frame (no more than 12 hours)
Measure: Median (Inter-Quartile Range); unit: number of treatments
Arm/Group | Control - Jet Nebulizer | Study - Vibrating Mesh Nebulizer
Number analyzed (Participants) | 109 | 108
number of treatments | 3.0 [2.0 to 5.0] | 2 [1.0 to 3.0]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over treatment period ranging from 1 to 3 hours
Arm/Group | Control - Jet Nebulizer | Study - Vibrating Mesh Nebulizer
All-Cause Mortality (participants affected / at risk) | 0/109 | 0/108
Serious Adverse Events (participants affected / at risk) | 0/109 | 0/108
Other Adverse Events (participants affected / at risk) | 0/109 | 0/108

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-02-15): https://cdn.clinicaltrials.gov/large-docs/41/NCT02774941/Prot_SAP_ICF_000.pdf